CLINICAL TRIAL: NCT04637321
Title: Everyone Poops: An Evaluation of the Incidence and Risk Factors for Clostridioides Difficle Infection in Solid Organ Transplant Recipients
Brief Title: The Incidence and Risk Factors for Clostridioides Difficle Infection in Solid Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 059.PHA.2019.D
Record Dates: First submitted 2019-11-04; First posted 2020-11-19 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Infection in Solid Organ Transplant Recipients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Solid organ transplant — Data will be collected on all liver, kidney, pancreas and combined transplant recipients who received their graft(s) from April 1, 2015 to July 31, 2018

SUMMARY:
2.1. Study Objectives

* Primary Objective(s)
* Identify the incidence and risk of CDI within one year after kidney, liver, and/or pancreas transplant
* Secondary Objective(s)
* Identify the risk factors for recurrent CDI post-transplant in patients who were diagnosed with a CDI within one year prior to Solid Organ Transplant
* Evaluate the impact of CDI on graft survival following Solid Organ Transplant

DETAILED DESCRIPTION:
* Single center, retrospective cohort chart review study design
* Data will be collected on all liver, kidney, pancreas and combined transplant recipients who received their graft(s) from April 1, 2015 to July 31, 2018
* Will analyze outcomes from April 1, 2014 to July 31, 2019
* Patient list will be generated in Epic and Meditech
* All data will be obtained from Epic and Meditech
* All data will be collected retrospectively after the patient is discharged from the hospital

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant patients who received graft(s) at MDMC from April 1, 2015 to July 31, 2018
* Age >18 years old

Exclusion Criteria:

* Age <18 years old
* Loss to early death defined as within one week from transplantation
* Patients whose primary address is in Puerto Rico

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant patients who received graft(s) at MDMC from April 1, 2015 to July 31, 2018
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence of C. Difficile infection (CDI) within one year post-transplant | April 1, 2014 to July 31, 2019
  Incidence of C. Difficile infection within one year post-transplant for CDI post-transplant.
Risk factors for CDI post-transplant - No.1 | April 1, 2014 to July 31, 2019
  Risk factors transplanted organ
Risk factors for CDI post-transplant - No.2 | April 1, 2014 to July 31, 2019
  Origin of transplanted graft including age of donor
Risk factors for CDI post-transplant No.-3 | April 1, 2014 to July 31, 2019
  Induction agent used
Risk factors for CDI post-transplant No.4 | April 1, 2014 to July 31, 2019
  Acid suppression
Risk factors for CDI post-transplant No.5 | April 1, 2014 to July 31, 2019
  First time SOT recipient
Risk factors for CDI post-transplant No.6 | April 1, 2014 to July 31, 2019
  History of CDI in the year prior to transplant
Risk factors for CDI post-transplant No.7 | April 1, 2014 to July 31, 2019
  Co-infection with HIV/AIDS
Risk factors for CDI post-transplant No.8 | April 1, 2014 to July 31, 2019
  Length of hospital stay
Risk factors for CDI post-transplant No. 9 | April 1, 2014 to July 31, 2019
  Length of intensive care unit stay
Risk factors for CDI post-transplant No.10 | April 1, 2014 to July 31, 2019
  Intra-operative administration of blood products
Risk factors for CDI post-transplant No. 11 | April 1, 2014 to July 31, 2019
  Antibiotic use in the 90 days prior to infection
Risk factors for CDI post-transplant No. 12 | April 1, 2014 to July 31, 2019
  Antibiotic use in the 90 days post-transplant
Risk factors for CDI post-transplant No, 13 | April 1, 2014 to July 31, 2019
  Hospitalization in the 90 days prior to transplantation
Risk factors for CDI post-transplant No, 14 | April 1, 2014 to July 31, 2019
  Hospitalization in the 90 days post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Crotty, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Jessica Rago, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided